CLINICAL TRIAL: NCT05196373
Title: A Phase I/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity and Preliminary Efficacy of STP705 Administered as Intrascar Injection in Adult Patients With Hypertrophic Scars
Brief Title: Safety, Tolerability, Pharmacokinetics, Immunogenicity and Efficacy of STP705 in Adult Patients With Hypertrophic Scars
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sirnaomics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SRN-705-009
Record Dates: First submitted 2021-12-15; First posted 2022-01-19 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Hypertrophic Scar
MeSH Terms: conditions — Cicatrix, Hypertrophic

STUDY DESIGN:
Intervention Model Description: Open label, Dose Escalation and Dose Expansion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Part 1: Group 1 (Experimental): 10ug Intrascar injection
  Interventions: Drug: STP705
- Part 1: Group 2 (Experimental): 20ug Intrascar injection
  Interventions: Drug: STP705
- Part 1: Group 3 (Experimental): 40ug Intrascar injection
  Interventions: Drug: STP705
- Part 1: Group 4 (Experimental): 60ug Intrascar injection
  Interventions: Drug: STP705
- Part 1: Group 5 (Experimental): 80ug Intrascar injection
  Interventions: Drug: STP705
- Part 1: Group 6 (Experimental): 100ug Intrascar injection
  Interventions: Drug: STP705

INTERVENTIONS:
Drug: STP705 — STP705 Powder for Injection composed of siRNA-TGF-B1 and siRNA-COX-2 packged in a proprietary polymer nanoparticle formulation for delivery.

SUMMARY:
Adult patients with hypertrophic scars 30 Subjects in Dose Escalation 20 Subjects in Dose Expansion Intrascar injection of STP705 weekly for 4 weeks

DETAILED DESCRIPTION:
An open label study design to evaluate the preliminary efficacy of STP705 in adult patients with hypertrophic scars.

The study is divided into 2 stages:

1. Dose Escalation: 30 subjects to be enrolled in this stage with a total of 6 dose groups.

3 subjects will be enrolled in 10ug and 20ug groups and 6 subjects in the subsequent groups of 40ug, 60ug, 80u and 100ug.

2. Dose Expansion:1-2 dose groups will be selected and 20 subjects will be enrolled in each group.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult ≥ 18 and ≤ 45 years old at the time of signing the ICF,
2. Diagnosed with hypertrophic scars, with all the following characteristics:

   1. Linear hypertrophic scar, with a width of 0.3-1.0 cm and a length of ≥10 cm;
   2. Scars with any of the following characteristics: redness or purpleness, stiffness, rough surface, significant swelling, visible dilated capillaries on the surface, and possibly accompanied by pain or itching;
   3. The course of the disease is 6 to 24 months (inclusive);
   4. Scars are not located on the face, front of the neck, feet, hands, knees, elbows or any joints;
3. The examination during the screening period must meet the following criteria: medical history, physical examination (excluding hypertrophic scar), 12-lead ECG, vital signs, laboratory examinations are judged by the investigator to meet the requirements, and no clinically significant abnormalities were observed;
4. Subjects of childbearing potential (male or female) must take effective medical contraceptive measures during the study and within 6 months after the end of administration;
5. Subjects voluntarily participate in this clinical trial and sign the ICF, can understand and comply with the study procedures, and complete the entire study as specified by the protocol.

Exclusion Criteria:

1. Diagnosed with keloid or burn scar;
2. Positive in hepatitis B surface antigen, hepatitis C antibody, human immunodeficiency virus (HIV), or syphilis antibody tests;
3. Medication history of corticosteroids use (including inhaled steroids, triamcinolone acetonide, etc.) and COX-2 inhibitors within 3 months before the first injection of the study (if 5 times the half-life is longer than 3 months, then 5 times the half-life will prevail);
4. Impaired immune function (such as cancer, or other diseases that affect the basic immune responses);
5. Concomitant diseases that is uncontrolled or poorly controlled or may affect the study, including clinically important cardiovascular, lung, kidney, endocrine, liver, nerve, mental, immune, gastrointestinal, blood, urogenital, skeletal or metabolic disorders at the investigator's discretion;
6. Known to be allergic to STP705 or any components of its prescription;
7. Having difficulty in venous blood collection, or having a history of needle fainting or blood fainting;
8. Infection or trauma in the site to be treated;
9. Pregnant and lactating women;
10. Participated in other clinical studies and received treatment within 3 months before the first injection;
11. Blood donation or blood loss ≥400 mL within 3 months before the first injection (except for female blood loss during menstrual period), or planning to donate blood or blood components during the study period or within 3 months after the end of the study;
12. History of drug abuse/dependence or drug history or positive in drug abuse screening (screening items can include: morphine, tetrahydrocannabinol acid, methamphetamine, methylenedioxy methanphetamine, ketamine and cocaine) within 1 year before the first injection;
13. Medication history of any drugs (including prescription drugs, over-the-counter drugs, Chinese herbal medicines, etc.) or health care products within 14 days before the first injection;
14. Vaccinated with live vaccines within 4 weeks before the first injection or planning to receive live vaccines within 4 weeks after the last dose. Live vaccines include but not limited to: measles, mumps, rubella, chickenpox, yellow fever, rabies, Bacillus Calmette-Guerin, typhoid fever, COVID-19 live vaccines, etc.;
15. Any surgical, medical or laboratory pathophysiological conditions that may interfere with the safety, distribution, metabolism or excretion of the investigational drug at the discretion of the investigator;
16. Unable to communicate or cooperate with medical staff due to neurological, mental disorders or language/ verbal communication issues;
17. Other situations not suitable for participation in the study as judged by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Concentration of siRNA-TGF-B1 and siRNA-COX-2 in serum | 7 weeks
  siRNA-TGF-B1 and siRNA-COX-2 and HKP will be calculated

SECONDARY OUTCOMES:
Change of the scar from baseline using Observer Scar Assessment Scale | 7 weeks
  The scale will be used to record: vascularity, pigmentation, thickness, releif, pliability, surface area of the scar where 1= Normal skin and 10 = the worst case.
Change of the scar from baseline using Patient scale | 7 weeks
  The scale will be used to record: pain, itching, color, hardness, thickness, and relief where 1= No, not different from normal and 10 = Yes, very different from normal.

IPD SHARING:
Plan to Share IPD: Undecided